CLINICAL TRIAL: NCT02477436
Title: A Randomized, Placebo Controlled, Double Blind, Multicenter Therapeutic Exploratory Clinical Study for the Evaluation of the Efficacy and Safety of Avanafil in the Patients With Erectile Dysfunction
Brief Title: Efficacy and Safety of Avanafil in the Patients With Erectile Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Avanafil-Korea
Record Dates: First submitted 2015-06-03; First posted 2015-06-22 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — avanafil; Phosphodiesterase 5 Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Avanafil 50mg group (Experimental): Avanafil 50mg tablet + Placebo 100mg tablet
  Interventions: Drug: Avanafil
- Avanafil 100mg group (Experimental): Avanafil 100mg tablet + Placebo 100mg tablet
  Interventions: Drug: Avanafil
- Avanafil 200mg group (Experimental): Avanafil 100mg 2 tablets
  Interventions: Drug: Avanafil
- Placebo group (Placebo Comparator): Placebo 100mg 2tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avanafil — * One capsule should be taken with water, 30 minutes before sexual intercourse. It should be taken only once a day.
  * Intemperance in eating and drinking should not be done, 2 hours before and 2 hour after taking the investigational product.
  * Investigational products were administered prior to the sexual intercourse for total 8 weeks.
  Other Names: Phosphodiesterase 5 inhibitor
  Arms: Avanafil 100mg group; Avanafil 200mg group; Avanafil 50mg group
Drug: Placebo — * One capsule should be taken with water, 30 minutes before sexual intercourse. It should be taken only once a day.
  * Intemperance in eating and drinking should not be done, 2 hours before and 2 hour after taking the placebo.
  * Placebos were administered prior to the sexual intercourse for total 8 weeks.
  Arms: Placebo group

SUMMARY:
This is an exploratory clinical study to presume the optimum usage and dosage for a therapeutic confirmatory study by evaluating the efficacy and safety of Avanafil 50mg, 100mg, 200mg or placebo administered orally in patients with erectile dysfunction. In conclusions, Patients with erectile dysfunction (ED) were administered placebo, Avanafil 50mg, 100mg or 200mg 30 minutes before sexual intercourse for 8 weeks.

DETAILED DESCRIPTION:
1. Study design: Prospective, randomized, double blind, placebo-controlled, therapeutic exploratory clinical study Usage & period One capsule was administered 30minutes before sexual intercourse.It was administered only once a day.

[Evaluation endpoints]

1. Safety: ① Laboratory tests: Hematological Test, Blood chemical Test, Urinalysis Vital signs: blood pressure, pulse rate ③ Adverse events and Adverse drug reaction ④12-lead ECG
2. Efficacy

   * Primary endpoint ▪ The change of erectile function (EF) domain score in the international index of erectile function (IIEF)
   * Secondary endpoint ▪ The change of success rate in sexual encounter profile (SEP) questionnaire 2, questionnaire 3, questionnaire 4 and questionnaire 5 ▪ The change of score in IIEF questionnaire 3 and questionnaire 4, The change of score in other domains of IIEF, GEAQ (Global efficacy assessment question), Normal erectile function (IIEF EF domain score ≥ 26) rate Statistical methods

     1. Definition of Evaluation population Maximum efficacy evaluation population included the subjects who satisfied inclusion criteria, who took the investigational product at least once, who visited the hospital after taking the investigational product, and who got the result of efficacy evaluation. Safety-Evaluation Population consisted of the subjects who made a visit after taking the investigational product once or more and who got follow-up safety results
     2. Initial Comparability Discrete variables were comparatively analyzed by χ2-test, Fisher's exact test, and Successive variables were comparatively analyzed by ANOVA test or Kruskal-Wallis test.
     3. Efficacy Evaluation The change of EF domain score in the IIEF: Analysis of covariance(ANCOVA), in which baseline was corrected, was performed to check whether there was a difference between the placebo group and the Avanafil groups in change of EF domain score.

        The change of score in other domains of IIEF: Analysis of covariance(ANCOVA), in which baseline was corrected, was performed to check whether there was a difference between the placebo group and the Avanafil groups.

        The change of score in IIEF questionnaire 3 and questionnaire 4: Analysis of covariance(ANCOVA), in which baseline was corrected, was performed to check whether there was a difference between the placebo group and the Avanafil groups in IIEF questionnaire 3, questionnaire 4 respectively.

        The change of success rate in SEP questionnaire 2, questionnaire 3, questionnaire 4 and questionnaire 5: Analysis of covariance(ANCOVA), in which baseline was corrected, was performed to check whether there was a difference between the placebo group and the Avanafil groups.

        GEAQ (Global Efficacy Assessment Question) : The difference of GEAQ between groups was analyzed by χ2-test.

        Normal erectile function(IIEF EF domain score ≥ 26) rate: The difference of Normal erectile function rate between groups was analyzed by χ2-test.

        The efficacy results were analyzed by Dunnett's or Bonferroni's multiple comparison test to check whether there was a significant difference between the placebo group and the Avanafil groups.
     4. Safety Evaluation Adverse Events and Adverse Drug Reaction: The difference between the placebo group and the Avanafil groups was compared by using χ2-test or Fisher's exact test. Adverse events reported in study subjects were presented by WHOART (World Health Organization Adverse Reaction Terminology) system organ class. The adverse drug reactions, related with the investigational product, were comparatively verified on the same method.

All statistical analyses were performed under significance level 5%, test power 80% and two-side test.

ELIGIBILITY:
Inclusion Criteria:

1. The male subjects who were aged 19 ~ 70 with history of erectile dysfunction for at least 6 months duration
2. The subjects who had had stable monogamous relationships with their female partners
3. Their partners were free from pregnancy and lactation and well prevent conception
4. The subjects who were judged to be suitable to the clinical study in consequence of screening test
5. The subjects who consented to participate in the clinical study in writing
6. The subjects who attempted sexual intercourses at least 4 times in separate days during 4 weeks' free run-in period, and whose failure rate was over 50%.
7. The subjects whose point were between 11 and 25 in EF domain of IIEF after 4 weeks' free run-in period

Exclusion Criteria:

The following cases were excluded from this clinical study.

1. The subjects who had spinal cord injury or who underwent radical prostatectomy
2. The subjects whose penises were anatomically deformed (Ex: server penile fibrosis, and Peyronie's disease)
3. The subjects who had erectile dysfunction due to neurogenic or endocrine cause (hyperprolactinemia, low serum testosterone levels, etc.)

   * Hyperprolactinemia: serum prolactin over 3 times higher than the upper limit
   * Low Testosterone: serum total testosterone less than the lower limit
4. The subjects who had uncontrolled major psychiatric disorder and did not accept therapies (includes major depressions and schizophrenia) or had significant neurological abnormalities (neurovascular disorder)
5. The subjects who underwent cancer chemotherapy within 1 year
6. The subjects who were addicted to alcohol or who had continuously misused dependent drugs
7. The subjects who had hepatic dysfunction or renal dysfunction as in the following:

   * Hepatic Dysfunction: GOT and GPT (glutamate-pyruvate transaminase) were three times higher than the upper limit
   * Renal Dysfunction: serum creatinine was over 2.0mg/dl
8. The subjects who had uncontrollable diabetes (FPG>180mg/dL)
9. The subjects who had proliferative diabetic retinopathy
10. The subjects who suffered from stroke, transient ischemic attacks, myocardial infarction, heart failure that needed to be medically treated, unstable angina or fatal arrhythmia or who underwent coronary artery bypass graft within 6 months
11. The subjects had serious hypotension (SBP/DBP(diastolic blood pressure) is less than 90/50mmHg in a sitting posture) or uncontrollable severe hypertension (SBP/DBP is over 170/100mmHg in a sitting posture)
12. The subjects who had hematological disorders that was likely to be developed into priapism such as sickle cell disease, multiple myeloma, leukemia
13. The subjects who had retinitis pigmentosa
14. The subjects who suffered from serious GI bleeding disorder within 1 year
15. The subjects who took Viagra®, Cialis®, Levitra®, Mvix® and others within 2 weeks before the clinical study
16. The subjects who had taken the following drugs

    ① Nitrate/Nitric oxide(NO) donors(ex. Nitroglycerin, isosorbide mononitrate, amyl nitrate/nitrite, sodium nitroprusside)

    ② Androgens(ex testosterone), anti-androgen, trazodone

    ③ Anticoagulant (excludes antiplatelet drugs)

    ④ Erythromycin, itraconazole, ketoconazole, cimetidine, ritonavir, saquinavir, amprenavir, indinavir and nelfinavir that greatly affects CYP3A4 (cytochrome P450 isoenzyme 3A4)
17. The subjects who had history of hypersensitivity to the PDE(phosphodiesterase)-5 inhibitors or whose erectile dysfunction was not improved
18. The subjects who had hypoactive sexual desire
19. The subjects who had no intention of having sexual intercourses 4 times in separate days during 4 weeks' free run-in period
20. The subjects who took other study drugs within 30 days before this clinical study
21. The subjects who were judged to be unsuitable to the clinical study by other reasons

Ages: 19 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change of erectile (EF) domain score in the international index of erectile function (IIEF) questionnaire | Week 4 and 8

SECONDARY OUTCOMES:
The change of success rate for SEP (Sexual encounter profile) questionnaire 2,3,4 and 5 | Week 4 and 8
The change of score in orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction domains in international index of erectile function (IIEF) | Week 4 and 8
The change of score in the international index of erectile function (IIEF) questionnaire 3 and 4 | Week 4 and 8
Improvement of erection on the GEAQ (Global Efficacy Assessment Question) questionnaire | Week 4 and 8
  The GEAQ question, 'Has the treatment you have been over the past 8weeks improved your erections?'
Normal erectile function (IIEF EF domain score ≥ 26) rate | Week 4 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Jun Park, PhD, MD, Principal Investigator — Department of Urology, Pusan National University Hospital
Locations (1):
- Department of Urology, Pusan National University Hospital, Busan, South Korea

REFERENCES:
- [Derived] Park HJ, Kim SW, Kim JJ, Lee SW, Paick JS, Ahn TY, Park K, Park JK, Park NC. A Randomized, Placebo-Controlled, Double-Blind, Multi-Center Therapeutic Confirmatory Study to Evaluate the Safety and Efficacy of Avanafil in Korean Patients with Erectile Dysfunction. J Korean Med Sci. 2017 Jun;32(6):1016-1023. doi: 10.3346/jkms.2017.32.6.1016. PMID 28480661